CLINICAL TRIAL: NCT01976416
Title: Novel Use Of Hydroxyurea in an African Region With Malaria
Acronym: NOHARM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Doris Duke Charitable Foundation (Other); Makerere University (Other); Mulago Hospital, Uganda (Other); Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Chandy John, Professor of Pediatrics, Medicine, Microbiology and Immunology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012139
Record Dates: First submitted 2013-10-22; First posted 2013-11-05 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Sickle Cell Anemia; Sickle Cell Disease; Malaria
Keywords: Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell; Malaria | interventions — Hydroxyurea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydroxyurea (Experimental): Fixed dose 20 ± 2.5 mg/kg/day, administered once a day in tablet form (100mg or scored 1000mg) for twelve months
  Interventions: Drug: Hydroxyurea
- Placebo (Placebo Comparator): Fixed dose 20 ± 2.5 mg/kg/day, administered once a day in tablet form (100mg or scored 1000mg) for twelve months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxyurea
  Other Names: Siklos; Hydroxycarbamide
  Arms: Hydroxyurea
Drug: Placebo
  Arms: Placebo

SUMMARY:
Multiple studies have shown that hydroxyurea has clinical efficacy in preventing acute painful episodes and reducing the need for blood transfusions in children with sickle cell anemia (SCA), but no study has been conducted in malaria endemic regions of sub-Saharan Africa, the areas with the most children with SCA.

The primary goal of this study is to investigate the safety and efficacy of hydroxyurea for children with SCA in a malaria endemic region within sub-Saharan Africa.

DETAILED DESCRIPTION:
The risk of malaria and hematologic toxicities from hydroxyurea in children with SCA living in malaria endemic regions is unknown.

Some changes associated with hydroxyurea treatment (increased nitric oxide and HbF) would be expected to protect against malaria, but the data on hydroxyurea-related endothelial changes thought to be important in malaria pathogenesis (e.g. intracellular adhesion molecule (ICAM)-1, von Willebrand factor (VWF), tumor necrosis factor (TNF)-α) is unclear, with some studies suggesting that these factors might be increased with hydroxyurea and others suggesting no difference or a decrease.

The specific aims of this study are as follows:

1. Determine the incidence of malaria in children with sickle cell anemia treated with hydroxyurea vs. placebo
2. Establish the frequency of hematologic toxicities and adverse events in children with sickle cell anemia treated with hydroxyurea vs. placebo
3. Define the relationship between hydroxyurea treatment and fetal hemoglobin (HbF), soluble ICAM-1 (sICAM-1) and nitric oxide (NO) levels, and between levels of these factors and risk of subsequent malaria.

Two hundred children from the Mulago Hospital Sickle Cell Clinic (MHSCC) in Kampala, Uganda will be randomized to receive either hydroxyurea (100) or placebo (100) at a fixed dose of 20 ± 2.5 mg/kg/day. The primary study endpoints will be evaluated after twelve months of study treatment. After twelve months of study treatment, children will enter a follow-up phase during which they can receive an additional twelve months of open-label hydroxyurea treatment if they/their parents wish to do so after consultation with local physicians at the MHSCC.

The working hypotheses of this research study are:

1. The incidence of malaria is not greater in children with SCA treated with hydroxyurea than those treated with placebo
2. Children with SCA treated with hydroxyurea will have more medication-related hematologic toxicities, such as neutropenia, but no increase in SCA-related adverse events (e.g. pain crises, hospitalizations, requirement for blood transfusion) compared to children treated with placebo
3. Hydroxyurea will increase HbF and plasma NO levels and decrease plasma sICAM-1 levels; HbF and plasma NO levels will inversely correlate, and plasma sICAM-1 levels will positively correlate, with subsequent malaria incidence

ELIGIBILITY:
Inclusion Criteria:

* Pediatric subjects with documented sickle cell anemia (HbSS supported by hemoglobin electrophoresis or by peripheral blood smear showing sickled red blood cells)
* Age range of 1.00-3.99 years, inclusive, at the time of enrollment
* Weight at least 5.0 kg at the time of enrollment
* Willingness to comply with all study-related treatments, evaluations, and follow up

Exclusion Criteria:

* Known chronic medical condition (e.g., HIV, malignancy, active clinical tuberculosis)
* Severe malnutrition determined by impaired growth parameters as defined by WHO (weight for length/height or weight-for-length/height > 3 z-scores below the median WHO growth standards)
* Pre-existing severe hematological toxicity:

  1. Hb <4.0 g/dL
  2. Hb <6.0 g/dL AND ARC <100 x 10E9/L
  3. Hb <7.0 g/dL AND ARC <80 x 10E9/L
  4. Platelets <80 x 10E9/L
  5. ANC <1.0 x 10E9/L
* Alanine transaminase (ALT) or creatinine >2 times the upper limit of normal for age
* Blood transfusion within 30 days prior to enrollment

Ages: 12 Months to 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 208 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandy C. John, M.D., Principal Investigator — Indiana University
Locations (1):
- Mulago Hospital Sickle Cell Clinic, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Opoka RO, Ndugwa CM, Latham TS, Lane A, Hume HA, Kasirye P, Hodges JS, Ware RE, John CC. Novel use Of Hydroxyurea in an African Region with Malaria (NOHARM): a trial for children with sickle cell anemia. Blood. 2017 Dec 14;130(24):2585-2593. doi: 10.1182/blood-2017-06-788935. Epub 2017 Oct 19. PMID 29051184
- [Derived] Power-Hays A, McElhinney KE, Williams TN, Mochamah G, Olupot-Olupot P, Paasi G, Reid ME, Rankine-Mullings AE, Opoka RO, John CC, McGann PT, Quinn CT, Punt NC, Smart LR, Stuber SE, Latham TS, Vinks AA, Ware RE. Hydroxyurea pharmacokinetics in children with sickle cell anemia across different global populations. Blood Adv. 2026 Jan 27;10(2):418-427. doi: 10.1182/bloodadvances.2025017254. PMID 41026975
- [Derived] Siegert TF, Opoka RO, Nakafeero M, Carman A, Mellencamp KA, Latham T, Hume H, Lane A, Ware RE, Ssenkusu JM, John CC, Conroy AL. Angiopoietin-2 is associated with sickle cell complications, including stroke risk, and decreases with hydroxyurea therapy. Blood Vessel Thromb Hemost. 2024 Feb 8;1(1):100001. doi: 10.1016/j.bvth.2024.100001. eCollection 2024 Mar. PMID 40765704
- [Derived] Carman AS, Sautter C, Anyanwu JN, Ssemata AS, Opoka RO, Ware RE, Rujumba J, John CC. Perceived benefits and risks of participation in a clinical trial for Ugandan children with sickle cell anemia. Pediatr Blood Cancer. 2020 Feb;67(2):e27830. doi: 10.1002/pbc.27830. Epub 2019 May 28. PMID 31135090
- [Derived] Anyanwu JN, Williams O, Sautter CL, Kasirye P, Hume H, Opoka RO, Latham T, Ndugwa C, Ware RE, John CC. Novel Use of Hydroxyurea in an African Region With Malaria: Protocol for a Randomized Controlled Clinical Trial. JMIR Res Protoc. 2016 Jun 23;5(2):e110. doi: 10.2196/resprot.5599. PMID 27339303

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydroxyurea: Fixed dose 20 ± 2.5 mg/kg/day, administered once a day in tablet form (100mg or scored 1000mg) for twelve months
  Hydroxyurea
- Placebo: Fixed dose 20 ± 2.5 mg/kg/day, administered once a day in tablet form (100mg or scored 1000mg) for twelve months
  Placebo
Period: Overall Study
Arm/Group | Hydroxyurea | Placebo
Started | 104 | 104
Completed | 102 | 102
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydroxyurea | Placebo | Total
Number analyzed (Participants) | 104 | 103 | 207
Age, Customized [Count of Participants; unit: Participants]
  Age 1.00-3.99 years | 104 | 103 | 207
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 46 | 95
  Male | 55 | 57 | 112
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Uganda | 104 | 103 | 207

OUTCOME MEASURES:

1. Primary Outcome: Number of Malaria Episodes
Description: Malaria is defined as the presence of P. falciparum or P. malariae on the peripheral smear of any child brought in for medical evaluation of fever. P. vivax, P. ovale and P. knowlesi are not known to be present in this region, but if a child is seen with suspected infection with any of these malaria parasites, this will also be recorded as a case of malaria. Incidence will be reported in the number of cases per 100 patient years.
Time Frame: 12 months
Measure: Number; unit: malaria episodes
Units Other Than Participants: person-years
Arm/Group | Hydroxyurea | Placebo
Number analyzed (Participants) | 104 | 103
Number analyzed (person-years) | 104 | 103
malaria episodes | 5 | 7

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Hydroxyurea | Placebo
All-Cause Mortality (participants affected / at risk) | 2/104 | 1/103
Serious Adverse Events (participants affected / at risk) | 6/104 | 6/103
Other Adverse Events (participants affected / at risk) | 76/104 | 88/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea (N=104) | Placebo (N=103)
Bacteremia (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Vaso-Occlusive Crisis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Splenic Squestration (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Sudden Death (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxyurea (N=104) | Placebo (N=103)
Vaso-Occlusive Crisis (Blood and lymphatic system disorders) | 38 (58) | 59 (106)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 21 (24) | 24 (32)
Clinical Sepsis (Infections and infestations) | 6 (8) | 13 (16)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 54 (107) | 62 (108)
Gastrointestinal-related (Gastrointestinal disorders) | 13 (15) | 12 (15)
Malaria (Blood and lymphatic system disorders) | 3 (5) | 7 (7)
Other infections (Infections and infestations) | 7 (8) | 14 (14)
Others (e.g., injury) (Injury, poisoning and procedural complications) | 7 (7) | 9 (10)
Anemia (Blood and lymphatic system disorders) | 25 (40) | 42 (65)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (12) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes